CLINICAL TRIAL: NCT01217957
Title: An Open-Label, Dose-Escalation, Phase 1/2 Study of the Oral Form of Ixazomib (MLN9708), a Second-Generation Proteasome Inhibitor, Administered in Combination With Lenalidomide and Low-Dose Dexamethasone in Patients With Newly Diagnosed Multiple Myeloma Requiring Systemic Treatment
Brief Title: A Study of Ixazomib Administered in Combination With Lenalidomide and Low-Dose Dexamethasone in Patients With Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C16005; U1111-1176-7340 (Registry Identifier: WHO)
Record Dates: First submitted 2010-09-24; First posted 2010-10-08 (Estimated); Results first posted 2016-01-27 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Multiple Myeloma
Keywords: Drug therapy
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Phase 1: Ixazomib 1.68 mg/m^2 + Lenalidomide + Dexamethasone (Experimental): In phase 1, ixazomib 1.68 mg/m^2, capsules, orally, once, on Days 1, 8 and 15; plus dexamethasone 40 mg, tablets, orally, once on Days 1, 8, 15 and 22; and lenalidomide 25 mg, capsules, orally, once on Days 1 through 21 of a 28-day cycle for up to 12 cycles. Cycle 13 and beyond, single agent ixazomib 1.68 mg/m^2, capsules, orally, once on Days 1, 8 and 15 of a 28-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Ixazomib; Drug: Lenalidomide; Drug: Dexamethasone
- Phase 1: Ixazomib 2.23 mg/m^2 + Lenalidomide + Dexamethasone (Experimental): In phase 1, ixazomib 2.23 mg/m^2, capsules, orally, once, on Days 1, 8 and 15; plus dexamethasone 40 mg, tablets, orally, once on Days 1, 8, 15 and 22; and lenalidomide 25 mg, capsules, orally, once on Days 1 through 21 of a 28-day cycle for up to 12 cycles. Cycle 13 and beyond, single agent ixazomib 2.23 mg/m^2, capsules, orally, once on Days 1, 8 and 15 of a 28-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Ixazomib; Drug: Lenalidomide; Drug: Dexamethasone
- Phase 1: Ixazomib 2.97 mg/m^2 + Lenalidomide + Dexamethasone (Experimental): In phase 1, ixazomib 2.97 mg/m^2, capsules, orally, once, on Days 1, 8 and 15; plus dexamethasone 40 mg, tablets, orally, once on Days 1, 8, 15 and 22; and lenalidomide 25 mg, capsules, orally, once on Days 1 through 21 of a 28-day cycle for up to 12 cycles. Cycle 13 and beyond, single agent ixazomib 2.97 mg/m^2, capsules, orally, once on Days 1, 8 and 15 of a 28-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Ixazomib; Drug: Lenalidomide; Drug: Dexamethasone
- Phase 1: Ixazomib 3.95 mg/m^2 + Lenalidomide + Dexamethasone (Experimental): In phase 1, ixazomib 3.95 mg/m^2, capsules, orally, once, on Days 1, 8 and 15; plus dexamethasone 40 mg, tablets, orally, once on Days 1, 8, 15 and 22; and lenalidomide 25 mg, capsules, orally, once on Days 1 through 21 of a 28-day cycle for up to 12 cycles. Cycle 13 and beyond, single agent ixazomib 3.95 mg/m^2, capsules, orally, once on Days 1, 8 and 15 of a 28-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Ixazomib; Drug: Lenalidomide; Drug: Dexamethasone
- Phase 2: Ixazomib 4.0 mg + Lenalidomide + Dexamethasone (Experimental): In phase 2, ixazomib 4.0 mg fixed dose, capsules, orally, once, on Days 1, 8 and 15; plus dexamethasone 40 mg, tablets, orally, once on Days 1, 8, 15 and 22; and lenalidomide 25 mg, capsules, orally, once on Days 1 through 21 of a 28-day cycle for up to 12 cycles. Cycle 13 and beyond, single agent ixazomib 4.0 mg fixed dose, capsules, orally, once on Days 1, 8 and 15 of a 28-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Ixazomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ixazomib — Ixazomib capsules
  Other Names: MLN9708; NINLARO®
Drug: Lenalidomide — Lenalidomide capsules
Drug: Dexamethasone — Dexamethasone tablets

SUMMARY:
The purpose of Phase 1 of this study was to determine the safety, tolerability, maximum tolerated dose (MTD), and recommended Phase 2 dose (RP2D) of oral ixazomib administered in combination with lenalidomide and low-dose dexamethasone in participants with newly diagnosed multiple myeloma (NDMM). The purpose of Phase 2 of this study was to determine the overall response rate (ORR) and further evaluate the tolerability and toxicity of the combination of oral ixazomib, lenalidomide, and low-dose dexamethasone in patients with NDMM.

DETAILED DESCRIPTION:
The drug being tested in this study is called ixazomib. Ixazomib was being tested to treat people who had newly diagnosed multiple myeloma who had not previously received systemic treatment. This study was conducted in two Phases. Phase 1 looked at side effects and lab results in people who took ixazomib to determine the MTD and RP2D. Phase 2 looked at overall response rates and side effects in people who took ixazomib.

The study enrolled 15 patients in Phase 1 and 50 patients in Phase 2. Participants in Phase 1 were assigned to cohorts and received ixazomib 1.68, 2.23, 2.97, or 3.95 mg/m^2 in addition to dexamethasone 40 mg and lenalidomide 25 mg. Participants in Phase 2 received ixazomib 4.0 mg fixed dose in addition to dexamethasone 40 mg and lenalidomide 25 mg. In both Phases study treatment was administered in 28-day Cycles as follows: ixazomib Days 1, 8 and 15, dexamethasone Days 1, 8, 15 and 22, and lenalidomide 25 mg Days 1 through 21.

This multi-center trial was conducted in the United States. The overall time to participate in this study was 12, 28-day cycles with the option to continue into a maintenance portion in the absence of disease progression or unacceptable toxicity. Participants made multiple visits to the clinic and a final visit 30 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following eligibility criteria to be enrolled in the study:

* Male or female patients 18 years or older
* Previously untreated multiple myeloma diagnosed according to standard criteria requiring systemic treatment
* Patients must have measurable disease
* Nonsecretory multiple myeloma based upon standard M-component criteria (i.e., measurable serum/urine M-component) is not allowed unless the baseline serum free light chain level (Freelite™) is evaluated Patients must meet clinical laboratory criteria as specified in study protocol
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Female and male patients MUST adhere to the guidelines of the lenalidomide pregnancy prevention program
* Must be able to take concurrent aspirin 325 mg daily
* Voluntary written consent

Exclusion Criteria

Patients meeting any of the following exclusion criteria are not to be enrolled in the study:

* Peripheral neuropathy that is greater or equal to Grade 2
* Female patients who are lactating or pregnant
* Major surgery or radiotherapy within 14 days before the first dose of study drug
* Serious infection requiring systemic antibiotic therapy within 14 days before the first dose of study drug
* Diarrhea greater than Grade 1 based on the National Cancer Institute Common Terminology Criteria for Adverse Events
* Central nervous system involvement.
* Evidence of current uncontrolled cardiovascular conditions within the past 6 months
* Known human immunodeficiency virus (HIV) positive, hepatitis B surface antigen-positive status, or known or suspected active hepatitis C infection
* Serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to the protocol
* Known gastrointestinal condition that could interfere with swallowing or the oral absorption or tolerance of ixazomib
* No other prior malignancy within 2 years except nonmelanoma skin cancer or carcinoma in situ of any type if they have undergone complete resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2010-11-22 (Actual); Primary Completion 2013-03-08 (Actual); Study Completion 2018-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (16):
- United States (16):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Cedars Sinai Medical Center, Los Angeles, California
  - Rocky Mountain Cancer Center Rose, Denver, Colorado
  - Cancer Center of Central Connecticut, Southington, Connecticut
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Mt Sinai Medical Center, Miami Beach, Florida
  - Emory University, Atlanta, Georgia
  - Harry and Jeannette Weinberg Cancer Center at Franklin Square Hospital, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - New York Presbyterian Hospital - Weill-Cornell, New York, New York
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - W VA University Mary Babb Randolph Cancer Center, Morgantown, West Virginia
  - The Medical College of Wisconsin, Inc., Milwaukee, Wisconsin

REFERENCES:
- [Derived] Gupta N, Yang H, Hanley MJ, Zhang S, Liu R, Kumar S, Richardson PG, Skacel T, Venkatakrishnan K. Dose and Schedule Selection of the Oral Proteasome Inhibitor Ixazomib in Relapsed/Refractory Multiple Myeloma: Clinical and Model-Based Analyses. Target Oncol. 2017 Oct;12(5):643-654. doi: 10.1007/s11523-017-0524-3. PMID 28803351
- [Derived] Kumar SK, Berdeja JG, Niesvizky R, Lonial S, Laubach JP, Hamadani M, Stewart AK, Hari P, Roy V, Vescio R, Kaufman JL, Berg D, Liao E, Di Bacco A, Estevam J, Gupta N, Hui AM, Rajkumar V, Richardson PG. Safety and tolerability of ixazomib, an oral proteasome inhibitor, in combination with lenalidomide and dexamethasone in patients with previously untreated multiple myeloma: an open-label phase 1/2 study. Lancet Oncol. 2014 Dec;15(13):1503-1512. doi: 10.1016/S1470-2045(14)71125-8. Epub 2014 Nov 14. PMID 25456369

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study at 10 investigative sites in the United States from 22 November 2010 to data cut-off 08 March 2013.
Pre-assignment Details: Participants with a diagnosis of multiple myeloma were enrolled in 1 of 4 dose-escalation cohorts ixazomib 1.68, 2.23, 2.97 or 3.95 mg/m^2 in combination with lenalidomide, and dexamethasone to establish maximum tolerated dose (MTD) and Recommended Phase 2 Dose (RP2D) in Phase 2. 65 participants were enrolled; 15 in phase 1 and 50 in phase 2.
Groups:
- Phase 2: Ixazomib 4.0 mg + Lenalidomide + Dexamethasone: In phase 2, ixazomib 4.0 mg fixed dose, capsules, orally, once, on Days 1, 8 and 15; plus dexamethasone 40 mg, tablets, orally, once on Days 1, 8, 15 and 22; and lenalidomide 25 mg, capsules, orally, once on Days 1 through 21 of a 28-day cycle. Cycle 13 and beyond, single agent ixazomib 4.0 mg fixed dose, capsules, orally, once on Days 1, 8 and 15 of a 28-day cycle until disease progression or unacceptable toxicity.
Period: Phase 1
Arm/Group | Phase 1: Ixazomib 1.68 mg/m^2 + Lenalidomide + Dexamethasone | Phase 1: Ixazomib 2.23 mg/m^2 + Lenalidomide + Dexamethasone | Phase 1: Ixazomib 2.97 mg/m^2 + Lenalidomide + Dexamethasone | Phase 1: Ixazomib 3.95 mg/m^2 + Lenalidomide + Dexamethasone | Phase 2: Ixazomib 4.0 mg + Lenalidomide + Dexamethasone
Started | 3 | 3 | 6 | 3 | 0
Completed | 2 | 3 | 5 | 2 | 0
Not Completed | 1 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Patient | 1 | 0 | 1 | 1 | 0
Period: Phase 2
Arm/Group | Phase 1: Ixazomib 1.68 mg/m^2 + Lenalidomide + Dexamethasone | Phase 1: Ixazomib 2.23 mg/m^2 + Lenalidomide + Dexamethasone | Phase 1: Ixazomib 2.97 mg/m^2 + Lenalidomide + Dexamethasone | Phase 1: Ixazomib 3.95 mg/m^2 + Lenalidomide + Dexamethasone | Phase 2: Ixazomib 4.0 mg + Lenalidomide + Dexamethasone
Started | 0 | 0 | 0 | 0 | 50
Completed | 0 | 0 | 0 | 0 | 49 (Completed=Participants who are ongoing or who have died on study.)
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Patient | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Population: all participants who received at least one dose of any of the 3 study drugs.
Groups:
- Phase 1 :Ixazomib 2.23 mg/m^2 + Lenalidomide + Dexamethasone: In phase 1, ixazomib 2.23 mg/m^2, capsules, orally, once, on Days 1, 8 and 15; plus dexamethasone 40 mg, tablets, orally, once on Days 1, 8, 15 and 22; and lenalidomide 25 mg, capsules, orally, once on Days 1 through 21 of a 28-day cycle for up to 12 cycles. Cycle 13 and beyond, single agent ixazomib 2.23 mg/m^2, capsules, orally, once on Days 1, 8 and 15 of a 28-day cycle until disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Phase 1: Ixazomib 1.68 mg/m^2 + Lenalidomide + Dexamethasone | Phase 1 :Ixazomib 2.23 mg/m^2 + Lenalidomide + Dexamethasone | Phase 1: Ixazomib 2.97 mg/m^2 + Lenalidomide + Dexamethasone | Phase 1: Ixazomib 3.95 mg/m^2 + Lenalidomide + Dexamethasone | Phase 2: Ixazomib 4.0 mg + Lenalidomide + Dexamethasone | Total
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 50 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (3.21) | 72.3 (4.51) | 63.2 (12.19) | 64.7 (9.29) | 64.2 (11.16) | 64.4 (10.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 3 | 2 | 20 | 29
  Male | 2 | 0 | 3 | 1 | 30 | 36
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 3 | 6 | 3 | 49 | 64
Race/Ethnicity, Customized [Number; unit: participants]
  White | 3 | 1 | 6 | 0 | 42 | 52
  Black or African American | 0 | 2 | 0 | 3 | 7 | 12
  Asian | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6 | 3 | 50 | 65
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6 | 3 | 50 | 65
Height [Mean (Standard Deviation); unit: cm] — Height data was available for 3, 3, 6, 3, 48 and 51 participants in each treatment arm, respectively.
  cm | 168.9 (12.90) | 155.4 (3.20) | 165.9 (10.21) | 171.1 (8.07) | 169.4 (11.57) | 168.5 (11.30)
Weight [Mean (Standard Deviation); unit: kg] | 87.43 (12.683) | 64.93 (16.045) | 72.82 (14.557) | 116.63 (25.480) | 86.13 (17.695) | 85.39 (19.247)
Body Surface Area [Mean (Standard Deviation); unit: m^2] — Body surface area is defined as [Height(cm) x Weight (kg)]/3600)^1/2. Body surface area data was available for 3, 3, 6, 3, 48 and 51 participants in each treatment arm, respectively.
  m^2 | 2.024 (0.2180) | 1.665 (0.1923) | 1.826 (0.2272) | 2.348 (0.3050) | 2.011 (0.2343) | 1.994 (0.2565)

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) as a Measure of Safety and Tolerability
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; or congenital anomaly; or a medically important event.
Time Frame: Until occurrence of progressive disease or unacceptable toxicity (Up to 336 days)
Population: The safety population was defined as all patients who received at least one dose of any of the 3 study drugs.
Measure: Number; unit: participants
Groups:
- Phase 1: Ixazomib 2.97 mg/m^2 + Lenalidomide + Dexamethasone: In phase 1, ixazomib 2.97 mg/m^2, capsules, orally, once, on Days 1, 8 and 15; plus dexamethasone 40 mg, tablets, orally, once on Days 1, 8, 15 and 22; and lenalidomide 25 mg, capsules, orally, once on Days 1 through 21 of a 28-day cycle. for up to 12 cycles. Cycle 13 and beyond, single agent ixazomib 2.97 mg/m^2, capsules, orally, once on Days 1, 8 and 15 of a 28-day cycle until disease progression or unacceptable toxicity.
Arm/Group | Phase 1: Ixazomib 1.68 mg/m^2 + Lenalidomide + Dexamethasone | Phase 1: Ixazomib 2.23 mg/m^2 + Lenalidomide + Dexamethasone | Phase 1: Ixazomib 2.97 mg/m^2 + Lenalidomide + Dexamethasone | Phase 1: Ixazomib 3.95 mg/m^2 + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 3 | 3 | 6 | 3
participants
  Any AE | 3 | 3 | 6 | 3
  SAE | 2 | 3 | 1 | 2

2. Primary Outcome: Phase 2: Objective Response Rate (ORR) Following Treatment With the Combination Of Oral Ixazomib, Lenalidomide And Low-Dose Dexamethasone
Description: ORR was defined as the percentage of participants with Complete (CR) + Very Good Partial Response (VGPR) assessed by the investigatory using International Myeloma Working Group (IMWG) Criteria. CR=Negative immunofixation on the serum and urine and; disappearance of any soft tissue plasmacytomas and; < 5% plasma cells in bone marrow. VGPR=Serum and urine M-protein detectable by immunofixation but not on electrophoresis or; 90% or greater reduction in serum M-protein plus urine M-protein level < 100 mg per 24 hours.
Time Frame: Until occurrence of progressive disease or unacceptable toxicity (Up to 787 days)
Population: Participants from the response-evaluable population, defined as all patients who received at least one dose of ixazomib, had measurable disease at baseline, and at least one post-baseline disease assessment, with available data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase 2: Ixazomib 4.0mg/2.23 + Lenalidomide + Dexamethasone: In phase 2, ixazomib 4.0 mg fixed dose, capsules, orally, once, on Days 1, 8 and 15; plus dexamethasone 40 mg, tablets, orally, once, on Days 1, 8, 15 and 22; and lenalidomide 25 mg, capsules, orally, once, on Days 1 through 21 of a 28-day cycle for up to 12 cycles. Cycle 13 and beyond, single agent ixazomib 4.0 mg fixed dose, capsules, orally, once on Days 1, 8 and 15 of a 28-day cycle until disease progression or unacceptable toxicity. Includes 3 participants who received 2.23. mg/m^2 in Phase 1.
Arm/Group | Phase 2: Ixazomib 4.0 mg + Lenalidomide + Dexamethasone | Phase 2: Ixazomib 4.0mg/2.23 + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 49 | 52
percentage of participants | 59 [44 to 73] | 62 [47 to 75]

3. Primary Outcome: Phase 1: Recommended Phase 2 Dose of Ixazomib Given in Combination With Lenalidomide and Low-Dose Dexamethasone
Description: RP2D will be determined based on number and type of adverse event and serious adverse events, assessments of clinical laboratory values, neurotoxicity grading, and treatment discontinuation.
Time Frame: Until occurrence of progressive disease or unacceptable toxicity (Up to 336 days)
Population: All Phase 1 participants.
Measure: Number; unit: mg/m^2
Groups:
- Phase 1: Ixazomib + Lenalidomide + Dexamethasone: In phase 1, ixazomib 1.68, 2.23, 2.97 or 3.95 mg/m^2, capsules, orally, once, on Days 1, 8 and 15; plus dexamethasone 40 mg, tablets, orally, once on Days 1, 8, 15 and 22; and lenalidomide 25 mg, capsules, orally, once on Days 1 through 21 of a 28-day cycle for up to 12 cycles. Cycle 13 and beyond, single agent ixazomib 1.68, 2.23, 2.97 or 3.95 mg/m^2, capsules, orally, once on Days 1, 8 and 15 of a 28-day cycle until disease progression or unacceptable toxicity.
Arm/Group | Phase 1: Ixazomib + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 15
mg/m^2 | 2.23

4. Primary Outcome: Phase 1: Maximum Tolerated Dose (MTD) of Ixazomib Administered Weekly in Combination With Lenalidomide and Low-Dose Dexamethasone
Description: MTD of ixazomib will be determined by assessing adverse events and serious adverse events, clinical laboratory values, neurotoxicity grading, and vital sign measurements.
Time Frame: Until occurrence of progressive disease or unacceptable toxicity (Up to 336 days)
Population: All Phase 1 participants.
Measure: Number; unit: mg/m^2
Arm/Group | Phase 1: Ixazomib + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 15
mg/m^2 | 2.97

5. Primary Outcome: Phase 2: Percentage of Participants With Grade 3 or Higher AEs, SAEs and Treatment Discontinuation
Description: as for outcome 1
Time Frame: Until occurrence of progressive disease or unacceptable toxicity (Up to 787 days)
Population: The safety population was defined as all patients who received at least one dose of any of the 3 study drugs.
Measure: Number; unit: percentage of participants
Groups:
- Phase 2 :Ixazomib 4.0 mg + Lenalidomide + Dexamethasone: In phase 2, ixazomib 4.0 mg fixed dose, capsules, orally, once, on Days 1, 8 and 15; plus dexamethasone 40 mg, tablets, orally, once on Days 1, 8, 15 and 22; and lenalidomide 25 mg, capsules, orally, once on Days 1 through 21 of a 28-day cycle for up to 12 cycles. Cycle 13 and beyond, single agent ixazomib 4.0 mg fixed dose, capsules, orally, once on Days 1, 8 and 15 of a 28-day cycle until disease progression or unacceptable toxicity.
- Phase 2: Ixazomib 4.0 mg/2.23 + Lenalidomide + Dexamethasone: In phase 2, ixazomib 4.0 mg fixed dose, capsules, orally, once, on Days 1, 8 and 15; plus dexamethasone 40 mg, tablets, orally, once, on Days 1, 8, 15 and 22; and lenalidomide 25 mg, capsules, orally, once, on Days 1 through 21 of a 28-day cycle for up to 12 cycles. Cycle 13 and beyond, single agent ixazomib 4.0 mg fixed dose, capsules, orally, once on Days 1, 8 and 15 of a 28-day cycle until disease progression or unacceptable toxicity. Includes 3 participants who received 2.23 mg/m^2 in Phase 1.
Arm/Group | Phase 2 :Ixazomib 4.0 mg + Lenalidomide + Dexamethasone | Phase 2: Ixazomib 4.0 mg/2.23 + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 50 | 53
percentage of participants
  Grade 3 or Higher AEs | 76 | 75
  SAEs | 40 | 43
  AEs Resulting in Treatment Discontinuation | 8 | 8

6. Secondary Outcome: Phase 1: Cmax: Maximum Observed Plasma Concentration for Ixazomib
Description: Cmax: Maximum Observed Plasma Concentration (Cmax) is the peak plasma concentration of ixazomib obtained directly from the plasma concentration-time curve.
Time Frame: Cycle 1, Days 1 and 15
Population: The Pharmacokinetic (PK) analysis population, defined as all patients enrolled in the phase 1 portion of the study who had sufficient dosing data and ixazomib concentration-time data to permit calculation of ixazomib pharmacokinetic parameters, with available data.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1: Ixazomib 1.68 mg/m^2 + Lenalidomide + Dexamethasone | Phase 1: Ixazomib 2.23 mg/m^2 + Lenalidomide + Dexamethasone | Phase 1: Ixazomib 2.97 mg/m^2 + Lenalidomide + Dexamethasone | Phase 1: Ixazomib 3.95 mg/m^2 + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 2 | 3 | 4 | 2
ng/mL
  Day 1 (n=1, 3, 4, 1) | NA (NA) — Not calculated for 1 participant. | 22.303 (13.0184) | 94.779 (34.5442) | NA (NA) — Not calculated for 1 participant.
  Day 15 (n=2, 3, 4, 1) | 11.999 (NA) — Not calculated for 2 participants. | 31.368 (31.9963) | 53.517 (22.1412) | NA (NA) — Not calculated for 1 participant.

7. Secondary Outcome: Phase 1: Tmax: Time to Reach the Maximum Observed Plasma Concentration (Cmax) for Ixazomib
Description: Tmax: Time to reach the first maximum observed plasma concentration (Cmax), equal to time (hours) to Cmax, obtained directly from the plasma concentration-time curve.
Time Frame: Cycle 1, Days 1 and 15
Population: The Pharmacokinetic (PK) analysis population, defined as all patients enrolled in the phase 1 portion of the study who had sufficient dosing data and ixazomib concentration-time data to permit calculation of ixazomib pharmacokinetic parameters, with data available.
Measure: Median (Full Range); unit: hours
Groups:
- Phase 1: Ixazomib 3.95 mg/m^2 + Lenalidomide + Dexamethasone: In phase 1, ixazomib 3.95 mg/m^2, capsules, orally, once, on Days 1, 8 and 15; plus dexamethasone 40 mg, tablets, orally, once on Days 1, 8, 15 and 22; and lenalidomide 25 mg, capsules, orally, once on Days 1 through 21 of a 28-day cycle up to 12 cycles. Cycle 13 and beyond, single agent ixazomib 3.95 mg/m^2, capsules, orally, once on Days 1, 8 and 15 of a 28-day cycle until disease progression or unacceptable toxicity.
Arm/Group | Phase 1: Ixazomib 1.68 mg/m^2 + Lenalidomide + Dexamethasone | Phase 1: Ixazomib 2.23 mg/m^2 + Lenalidomide + Dexamethasone | Phase 1: Ixazomib 2.97 mg/m^2 + Lenalidomide + Dexamethasone | Phase 1: Ixazomib 3.95 mg/m^2 + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 2 | 3 | 4 | 1
hours
  Day 1 (n=1, 3, 4, 1) | 1.020 [NA to NA] — Not calculated for 1 participant. | 1.520 [1.00 to 8.00] | 1.060 [0.50 to 1.08] | 0.250 [NA to NA] — Not calculated for 1 participant.
  Day 15 (n=2, 3, 4, 1) | 4.165 [1.05 to 7.28] | 1.000 [0.98 to 2.03] | 1.015 [1.00 to 2.02] | 2.000 [NA to NA] — Not calculated for 1 participant.

8. Secondary Outcome: Phase 1: AUC(0-168): Area Under the Plasma Concentration-Time Curve From Time 0 to 168 Hours Postdose for Ixazomib
Description: AUC(0-168) is a measure of the area under the plasma concentration-time curve from time 0 to 168 hours postdose for Ixazomib.
Time Frame: Cycle 1, Days 1 and 15
Population: as for outcome 6
Measure: Geometric Mean (Standard Deviation); unit: hr*ng/mL
Groups:
- Phase 1: Ixazomib 1.68 mg/m^2 + Lenalidomide + Dexamethasone: In phase 1, ixazomib 1.68 mg/m^2, capsules, orally, once, on Days 1, 8 and 15; plus dexamethasone 40 mg, tablets, orally, once on Days 1, 8, 15 and 22; and lenalidomide 25 mg, capsules, orally, once on Days 1 through 21 of a 28-day cycle up to 12 cycles. Cycle 13 and beyond, single agent ixazomib 1.68 mg/m^2, capsules, orally, once on Days 1, 8 and 15 of a 28-day cycle until disease progression or unacceptable toxicity.
- Phase 1: Ixazomib 2.23 mg/m^2 + Lenalidomide + Dexamethasone: In phase 1, ixazomib 2.23 mg/m^2, capsules, orally, once, on Days 1, 8 and 15; plus dexamethasone 40 mg, tablets, orally, once on Days 1, 8, 15 and 22; and lenalidomide 25 mg, capsules, orally, once on Days 1 through 21 of a 28-day cycle up to 12 cycles. Cycle 13 and beyond, single agent ixazomib 2.23 mg/m^2, capsules, orally, once on Days 1, 8 and 15 of a 28-day cycle until disease progression or unacceptable toxicity.
- Phase 1: Ixazomib 2.97 mg/m^2 + Lenalidomide + Dexamethasone: In phase 1, ixazomib 2.97 mg/m^2, capsules, orally, once, on Days 1, 8 and 15; plus dexamethasone 40 mg, tablets, orally, once on Days 1, 8, 15 and 22; and lenalidomide 25 mg, capsules, orally, once on Days 1 through 21 of a 28-day cycle up to 12 cycles. Cycle 13 and beyond, single agent ixazomib 2.97 mg/m^2, capsules, orally, once on Days 1, 8 and 15 of a 28-day cycle until disease progression or unacceptable toxicity.
Arm/Group | Phase 1: Ixazomib 1.68 mg/m^2 + Lenalidomide + Dexamethasone | Phase 1: Ixazomib 2.23 mg/m^2 + Lenalidomide + Dexamethasone | Phase 1: Ixazomib 2.97 mg/m^2 + Lenalidomide + Dexamethasone | Phase 1: Ixazomib 3.95 mg/m^2 + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 2 | 3 | 4 | 1
hr*ng/mL
  Day 1 (n=1, 3, 4, 1) | NA (NA) — Not calculated for 1 participant. | 587.667 (350.1861) | 923.484 (156.2679) | NA (NA) — Not calculated for 1 participant.
  Day 15 (n=2, 3, 3, 1) | 834.608 (NA) — Not calculated for 2 participants. | 1083.998 (104.0256) | 1831.324 (262.7420) | NA (NA) — Not calculated for 1 participant.

9. Secondary Outcome: Phase 1: Rac: Accumulation Ratio of Ixazomib
Description: The accumulation ratio (Rac) was estimated as the ratio of AUC(0-168) on Day 15 to the AUC(0-168) on Day 1. AUC(0-168) is the area under the plasma concentration-time curve from time 0 to 168 hours postdose for ixazomib.
Time Frame: Cycle 1, Day 15
Population: as for outcome 6
Measure: Geometric Mean (Standard Deviation); unit: Ratio
Arm/Group | Phase 1: Ixazomib 1.68 mg/m^2 + Lenalidomide + Dexamethasone | Phase 1: Ixazomib 2.23 mg/m^2 + Lenalidomide + Dexamethasone | Phase 1: Ixazomib 2.97 mg/m^2 + Lenalidomide + Dexamethasone | Phase 1: Ixazomib 3.95 mg/m^2 + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 1 | 3 | 3 | 0
Ratio | NA (NA) — Not calculated for 1 participant | 1.849 (0.8359) | 2.051 (0.6469) |

10. Secondary Outcome: Phase 1: Emax: Maximum Observed Inhibition of Whole Blood 20S Proteasome
Description: Emax is the maximum observed inhibition of whole blood 20S proteasome. The pharmacodynamics 20S Proteasome samples were collected and the assays were performed; however, concerns about the third-party laboratory's performance of the blood 20S proteasome activity assay were identified that precluded the ability to confirm the accuracy of the data so no data is reported.
Time Frame: Day 1 predose and at multiple time points (up to 168 hours) postdose and Day 15 predose and at multiple time points (up to 336 hours) postdose
Arm/Group | Phase 1: Ixazomib 1.68 mg/m^2 + Lenalidomide + Dexamethasone | Phase 1: Ixazomib 2.23 mg/m^2 + Lenalidomide + Dexamethasone | Phase 1: Ixazomib 2.97 mg/m^2 + Lenalidomide + Dexamethasone | Phase 1: Ixazomib 3.95 mg/m^2 + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Phase 1: TEmax: Time to the Maximum Observed Inhibition of Whole Blood 20S Proteasome
Description: TEmax is the time to the maximum observed inhibition of whole blood 20S proteasome. The pharmacodynamics 20S Proteasome samples were collected and the assays were performed; however, concerns about the third-party laboratory's performance of the blood 20S proteasome activity assay were identified that precluded the ability to confirm the accuracy of the data so no data is reported.
Time Frame: as for outcome 10
Arm/Group | Phase 1: Ixazomib 1.68 mg/m^2 + Lenalidomide + Dexamethasone | Phase 1: Ixazomib 2.23 mg/m^2 + Lenalidomide + Dexamethasone | Phase 1: Ixazomib 2.97 mg/m^2 + Lenalidomide + Dexamethasone | Phase 1: Ixazomib 3.95 mg/m^2 + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Phase 2: Time to Progression (TTP)
Description: TTP was measured as the time in months from the first dose of study treatment to the date of the first documented progressive disease (PD).
Time Frame: From the first dose of study treatment to the date of first documented progressive disease (Up to 787 days)
Population: The modified Intent-to-Treat (mITT) population was defined as all patients who received at least one dose of any study drug in phase 2 or who received at least one dose of any study drug and were treated at the phase 2 dose level during phase 1.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Phase 2: Ixazomib 4.0 mg/2.23 + Lenalidomide + Dexamethasone: In phase 2, ixazomib 4.0 mg fixed dose, capsules, orally, once, on Days 1, 8 and 15; plus dexamethasone 40 mg, tablets, orally, once, on Days 1, 8, 15 and 22; and lenalidomide 25 mg, capsules, orally, once, on Days 1 through 21 of a 28-day cycle for up to 12 cycles. Cycle 13 and beyond, single agent ixazomib 4.0 mg fixed dose capsules, orally, once on Days 1, 8 and 15 of a 28-day cycle until disease progression or unacceptable toxicity. Includes 3 participants who received 2.23 mg/m^2 in Phase 1.
Arm/Group | Phase 2: Ixazomib 4.0 mg + Lenalidomide + Dexamethasone | Phase 2: Ixazomib 4.0 mg/2.23 + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 50 | 53
months | NA [NA to NA] — Not estimable due to the low number of events. | NA [NA to NA] — Not estimable due to the low number of events.

13. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: OS was measured as the time in months from the first dose of study treatment to the date of death + 1 day.
Time Frame: From the first dose of study treatment to the date of death (up to 787 days)
Population: Safety Population included al participants who received 1 of the 3 study drugs. Participants who did not die were censored at the last study visit.
Measure: Median (95% Confidence Interval); unit: participants
Arm/Group | Phase 2: Ixazomib 4.0 mg + Lenalidomide + Dexamethasone | Phase 2: Ixazomib 4.0 mg/2.23 + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 50 | 53
participants | NA [NA to NA] — Not estimable due to the low number of participants who died. | NA [NA to NA] — Not estimable due to the low number of participants who died.

14. Secondary Outcome: Phase 2: Overall Response Rate (ORR)
Description: ORR was defined as the percentage of participants with CR, VGPR and Partial Response (PR) assessed by the investigator using IMWG criteria. CR=Negative immunofixation on the serum and urine + Disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow. PR=50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by 90% or to < 200 mg per 24 hours. VGPR= Serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level < 100 mg per 24 hours.
Time Frame: Up to 787 days
Population: The response-evaluable population was defined as all patients who received at least one dose of ixazomib, had measurable disease at baseline, and at least one post-baseline disease assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Ixazomib 4.0 mg + Lenalidomide + Dexamethasone | Phase 2: Ixazomib 4.0 mg/2.23 + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 49 | 52
percentage of participants | 88 [75 to 95] | 88 [77 to 96]

15. Secondary Outcome: Phase 2: Percentage of Participants With Complete Response (CR) and Very Good Partial Response (VGPR)
Description: Response was assessed by the investigator using International Myeloma Working Group (IMWG) Criteria. CR is defined as negative immunofixation on the serum and urine and; disappearance of any soft tissue plasmacytomas and; < 5% plasma cells in bone marrow. VGPR is defined as Serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level < 100 mg per 24 hours.
Time Frame: After Cycles 3, 6 and 9 (Up to 787 days)
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Ixazomib 4.0 mg + Lenalidomide + Dexamethasone | Phase 2: Ixazomib 4.0 mg/2.23 + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 49 | 52
percentage of participants
  After 3 cycles | 35 [22 to 50] | 37 [24 to 51]
  After 6 cycles | 47 [33 to 62] | 48 [34 to 62]
  After 9 cycles | 57 [42 to 71] | 58 [43 to 71]

16. Secondary Outcome: Phase 2: Percentage of Participants With Complete Response (CR), Stringent Complete Response (sCR), Very Good Partial Response (VGPR), Near Complete Response (nCR), Partial Response (PR) and Minimal Response (MR)
Description: Response was assessed by the investigator using International Myeloma Working Group (IMWG) Criteria. CR=Negative immunofixation on the serum and urine + Disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow. sCR= CR + Normal free light chain (FLC) ratio and Absence of clonal cells in bone marrow. PR=≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to < 200 mg per 24 hours. VGPR= Serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level < 100 mg per 24 hours. nCR=Positive immunofixation analysis of serum or urine as the only evidence of disease. Disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow. MR=25% to 49% reduction in serum paraprotein and 50% to 89% reduction in urine light chain excretion for 6 weeks.
Time Frame: Cycles 3, 6, 9 and 12 (Up to 787 days)
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Ixazomib 4.0 mg + Lenalidomide + Dexamethasone | Phase 2: Ixazomib 4.0 mg/2.23 + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 49 | 52
percentage of participants
  CR | 20 [10 to 34] | 23 [13 to 37]
  sCR | 6 [1 to 17] | 10 [3 to 21]
  VGPR | 39 [25 to 54] | 38 [25 to 53]
  nCR | 2 [NA to 11] — 95% CI lower limit is <1. | 2 [NA to 10] — 95% CI lower limit is <1.
  PR | 67 [52 to 80] | 65 [51 to 78]
  MR | 6 [1 to 17] | 6 [1 to 16]

17. Secondary Outcome: Phase 2: Time to Best Response
Description: Time to Best Response was measured as the time in months from the first dose of study treatment to the date of first documented documentation of a confirmed response of partial response (PR) or better.
Time Frame: Up to 787 days
Population: Participants form the response-evaluable population, defined as all patients who received at least one dose of ixazomib, had measurable disease at baseline, and at least one post-baseline disease assessment, with available data.
Measure: Median (Full Range); unit: months
Arm/Group | Phase 2: Ixazomib 4.0 mg + Lenalidomide + Dexamethasone | Phase 2: Ixazomib 4.0 mg/2.23 + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 43 | 46
months | 2.96 [0.9 to 11.3] | 3.01 [0.9 to 12.9]

18. Secondary Outcome: Phase 2: Duration of Response (DOR)
Description: DOR was measured as the time in months from the date of first documentation of a confirmed response (CR + PR+ VGPR) to the date of the first documented disease progression (PD). Response was assessed by the investigator using International Myeloma Working Group (IMWG) Criteria. CR=negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow. VGPR=Serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level < 100 mg per 24 hours.
Time Frame: Up to 787 days
Population: Participants from the Response Evaluable Population, defined as all patients who received at least one dose of ixazomib, had measurable disease at baseline, and at least one post-baseline disease assessment, with data available for analysis. Patients who did not experience PD were censored at the last response assessment that was SD or better.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Ixazomib 4.0 mg + Lenalidomide + Dexamethasone | Phase 2: Ixazomib 4.0 mg/2.23 + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 49 | 52
months | NA [NA to NA] — Not estimable due to the low number of participants with events (progressive disease). | NA [NA to NA] — Not estimable due to the low number of participants with events (progressive disease).

19. Secondary Outcome: Phase 2: Progression Free Survival (PFS)
Description: PFS was measured as the time in months from the first dose of study treatment to the date of the first documented PD or death.
Time Frame: Up to 787 days
Population: The mITT population was defined as all patients who received at least one dose of any study drug in phase 2 or who received at least one dose of any study drug and were treated at the phase 2 dose level during phase 1.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Ixazomib 4.0 mg + Lenalidomide + Dexamethasone | Phase 2: Ixazomib 4.0 mg/2.23 + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 50 | 53
months | 14.98 [13.37 to NA] — Not estimable due to the low number of participants with events. | NA [NA to NA] — Not estimable due to the low number of participants with events.

20. Secondary Outcome: Phase 2: 1 Year Survival Rate
Description: 1-year survival rate is defined as the percentage of participants still alive at year after the first dose of stud drug.
Time Frame: 1 year after first dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase 2: Ixazomib 4.0 mg + Lenalidomide + Dexamethasone: In phase 2, ixazomib 4.0 mg fixed dose, capsules, orally, once, on Days 1, 8 and 15; plus dexamethasone 40 mg, tablets, orally, once on Days 1, 8, 15 and 22; and lenalidomide 25 mg, capsules, orally, once on Days 1 through 21 of a 28-day cycle. for up to 12 cycles. Cycle 13 and beyond, single agent ixazomib 4.0 mg fixed dose, capsules, orally, once on Days 1, 8 and 15 of a 28-day cycle until disease progression or unacceptable toxicity.
- Phase 2: Ixazomib 4.0 mg/2.23 + Lenalidomide + Dexamethasone: In phase 2, ixazomib 4.0 mg fixed dose, capsules, orally, once, on Days 1, 8 and 15; plus dexamethasone 40 mg, tablets, orally, once, on Days 1, 8, 15 and 22; and lenalidomide 25 mg, capsules, orally, once, on Days 1 through 21 of a 28-day cycle. Includes 3 participants who received 2.23 mg/m^2 in Phase 1.
Arm/Group | Phase 2: Ixazomib 4.0 mg + Lenalidomide + Dexamethasone | Phase 2: Ixazomib 4.0 mg/2.23 + Lenalidomide + Dexamethasone
Number analyzed (Participants) | 42 | 45
percentage of participants | 92 [80 to 97] | 92 [81 to 97]

ADVERSE EVENTS:
Time Frame: Up to 787 days
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Phase 1: Ixazomib + Lenalidomide + Dexamethasone | Phase 2: Ixazomib 4.0 mg + Lenalidomide + Dexamethasone
Serious Adverse Events (participants affected / at risk) | 8/15 | 20/50
Other Adverse Events (participants affected / at risk) | 15/15 | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Ixazomib + Lenalidomide + Dexamethasone (N=15) | Phase 2: Ixazomib 4.0 mg + Lenalidomide + Dexamethasone (N=50)
Pneumonia (Infections and infestations) | 1 | 4
Diverticulitis (Infections and infestations) | 0 | 1
Bone abscess (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1 — One treatment-emergent death occurred in the Phase 2: Ixazomib 4 mg treatment arm and is related to the full regimen (lenalidomide, dexamethasone, and ixazomib).
Sepsis (Infections and infestations) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 1
Fatigue (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 2
Pyrexia (General disorders) | 1 | 0
Hernia obstructive (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1
Embolism (Vascular disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 — One treatment-emergent death occurred in the Phase 2: Ixazomib 4 mg treatment arm and is not related to study treatment.
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Ixazomib + Lenalidomide + Dexamethasone (N=15) | Phase 2: Ixazomib 4.0 mg + Lenalidomide + Dexamethasone (N=50)
Leukopenia (Blood and lymphatic system disorders) | 1 | 7
Lymphopenia (Blood and lymphatic system disorders) | 3 | 7
Neutropenia (Blood and lymphatic system disorders) | 2 | 16
Tachycardia (Cardiac disorders) | 1 | 5
Deafness (Ear and labyrinth disorders) | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 3
Dry eye (Eye disorders) | 0 | 4
Eye pain (Eye disorders) | 1 | 1
Vision blurred (Eye disorders) | 1 | 6
Visual impairment (Eye disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 3 | 5
Abdominal pain (Gastrointestinal disorders) | 1 | 4
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 4
Dyspepsia (Gastrointestinal disorders) | 1 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 2
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 4
Chest pain (General disorders) | 1 | 0
Irritability (General disorders) | 1 | 2
Local swelling (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 7
Pain (General disorders) | 0 | 4
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 1
Folliculitis (Infections and infestations) | 1 | 0
Fungal skin infection (Infections and infestations) | 1 | 1
Herpes simplex (Infections and infestations) | 1 | 0
Nasal vestibulitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2
Oral herpes (Infections and infestations) | 2 | 2
Rash pustular (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 7 | 16
Urinary tract infection (Infections and infestations) | 0 | 3
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 2
Sunburn (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 6
Aspartate aminotransferase increased (Investigations) | 0 | 4
Blood alkaline phosphatase increased (Investigations) | 1 | 4
Blood creatinine increased (Investigations) | 1 | 7
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 2 | 3
Weight increased (Investigations) | 2 | 7
Decreased appetite (Metabolism and nutrition disorders) | 4 | 6
Gout (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 9
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 6
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 5
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 9
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 11
Amnesia (Nervous system disorders) | 0 | 3
Dysgeusia (Nervous system disorders) | 3 | 11
Headache (Nervous system disorders) | 3 | 8
Hypoaesthesia (Nervous system disorders) | 3 | 3
Memory impairment (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 5
Sinus headache (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 5
Agitation (Psychiatric disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 3
Insomnia (Psychiatric disorders) | 3 | 18
Mental status changes (Psychiatric disorders) | 1 | 1
Mood swings (Psychiatric disorders) | 1 | 0
Lower urinary tract symptoms (Renal and urinary disorders) | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Breast tenderness (Reproductive system and breast disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 14
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 4
Erythema (Skin and subcutaneous tissue disorders) | 1 | 3
Macule (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 3
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 4
Rash erythematous (Skin and subcutaneous tissue disorders) | 3 | 4
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 10
Rash papular (Skin and subcutaneous tissue disorders) | 2 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 6
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 3
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Hypertension (Vascular disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.